CLINICAL TRIAL: NCT00976066
Title: An Open-label, Non-randomized [11C]Carfentanil PET Study in Healthy Male Subjects to Investigate Brain Mu-opioid Receptor Occupancy, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of GSK1521498 and Naltrexone.
Brief Title: [11C]Carfentanil PET Study of GSK1521498
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 111848
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Obesity; Naltrexone; Carfentanil; Receptor Occupancy; mu-opioid Receptor; PET (Positron Emission Tomography); BOLD-fMRI
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1521498 (Experimental): Subjects will receive a dose of the experimental compound GSK1521498
  Interventions: Drug: Part A Assessing GSK1521498; Drug: Part B Assessing GSK1521498
- Naltrexone (Active Comparator): Subjects will receive a dose of the licensed pharmaceutical product, Naltrexone
  Interventions: Drug: Part C Assessing Naltrexone

INTERVENTIONS:
Drug: Part A Assessing GSK1521498 — Each participant will receive up to three [11C]carfentanil PET scans and up to two doses of GSK1521498 in total. The doses used will span the expected receptor occupancy range providing these were well tolerated in the first-time in human study.
  Each subject will receive baseline [11C]carfentanil PET and fMRI scans (PET Scan 1 and fMRI Scan 1, respectively), followed by two treatment sessions (Treatment Sessions 1 and 2). Treatment session 1 and 2 are followed by PET scans and an fMRI scan (session 1 only). Sessions will be separated by at least 12 days. PET scans will be timed to coincide with peak brain occupancy. fMRI will begin approximately 30-60 minutes after completion of the PET scan.
  Arms: GSK1521498
Drug: Part B Assessing GSK1521498 — The purpose of Part B is to establish the timecourse of receptor occupancy of GSK1521498. Each participant in Part B will receive up to three [11C]carfentanil PET scans and one single oral dose of GSK1521498 expected to provide 50-75% receptor occupancy (selected with reference to data from Part A).
  Each Part B subject will receive baseline [11C]carfentanil PET and fMRI scans (PET Scan 1 and fMRI Scan 1, respectively) followed by a single treatment session. The treatment session will consist of a single oral dose of GSK1521498 followed by two subsequent PET scans (PET Scans 2 and 3) and one fMRI scan (fMRI Scan 2).
  Arms: GSK1521498
Drug: Part C Assessing Naltrexone — A range of doses of naltrexone will be tested in up to 12 participants in an adaptive design. Each Part C participant will receive up to three [11C]carfentanil PET scans and a single oral dose of naltrexone. No dose of naltrexone will exceed 50 mg, the dose usually used therapeutically in the treatment of opiate and alcohol dependence. Each Part C subject will receive baseline [11C]carfentanil PET and fMRI scans (PET Scan 1 and fMRI Scan 1, respectively) followed by a single treatment session. The treatment session will consist of a single oral dose of naltrexone followed by two subsequent PET scans (PET Scans 2 and 3) and one fMRI scan (fMRI Scan 2).
  Arms: Naltrexone

SUMMARY:
The purpose of this study is to determine whether GSK1521498 attaches to sites in the brain called mu-opioid receptors that are involved in the liking reactions to palatable high fat and high sugar foods. We hope that blocking these receptors may modify certain behaviours that may lead to obesity.

DETAILED DESCRIPTION:
This imaging study will be an open-label, non-randomised PET receptor occupancy study in healthy male volunteers. The degree and time course of μ-opioid receptor occupancy (RO) following single oral doses of GSK1521498 will be estimated by [11C]carfentanil displacement. Previous pre-clinical and human PET studies indicate that [11C]carfentanil is selective for the μ-opioid receptor and can be used to estimate μ-opioid receptor occupancy in vivo.

The PK/PD relationship between plasma concentrations of GSK1521498 and μ-opioid RO will be described. Potential relationships between μ-opioid RO and functional magnetic resonance imaging (fMRI) endpoints, measured in a food reward paradigm, will be assessed as an exploratory aim. Additionally, the PK/PD relationships between plasma concentrations of naltrexone (a generic μ-opioid receptor antagonist), μ-opioid receptor occupancy, and fMRI measures of reward processing will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 25 and 65 years old inclusive.
* Body weight ≥ 50 kg and BMI within the range 18.5.0 - 30.0 kg/m2 (inclusive).
* Normal ECG.
* The subject is able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject.
* Compliance with birth control methods as described in the study protocol.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* The subject has a positive pre-study drug/alcohol screen.
* History of hepatitis B and /or C
* A positive result for an HIV test.
* Abnormal thyroid function
* Positive evaluation for depression.
* History of heavy alcohol use as described in the study protocol.
* The subject has participated in a clinical trial and has received an investigational product within: 90 days.
* Participation in other drug studies within a calendar year.
* Use of prohibited medications as described in the study protocol.
* History of sensitivity to any of the study medications.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Past or present use of tobacco products.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Previous radiation dosages in excess of levels acceptable to take part in this study.
* History of claustrophobia or history of neurological conditions.
* Presence of a cardiac pacemaker.
* Works as a welder, metal worker or machinist

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06-15 (Actual); Primary Completion 2009-12-07 (Actual); Study Completion 2009-12-07 (Actual)

PRIMARY OUTCOMES:
The degree and time-course of mu-opioid receptor occupancy by GSK1521498 in brain regions of interest as measured by PET | Assessed at various endpoints to be determined based on emerging results
The relationship between plasma concentration and mu-opioid receptor occupancy by GSK1521498 | Assessed at various endpoints to be determined based on emerging results

SECONDARY OUTCOMES:
Adverse events and clinically relevant changes in electrocardiography (ECG); vital signs (blood pressure, heart rate); POMS, Bond and Lader VAS, laboratory safety data and physical examination | Duration of study
Pharmacokinetic endpoints will be: AUC(0-∞), AUC(0-t), maximum observed plasma drug concentration (Cmax), time to maximum observed plasma drug concentration (Tmax), terminal elimination half-life (t½). | PK samples will be collected throughout the study
The degree and time-course of mu-opioid receptor occupancy by naltrexone in brain regions of interest as measured by PET | Assessed at various endpoints to be determined based on emerging results
The relationship between mu-opioid receptor occupancy by GSK1521498 and naltrexone and fMRI responses during expectation and receipt of a pleasant tasting reward (juice) | During fMRI scanning sessions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Rabiner EA, Beaver J, Makwana A, Searle G, Long C, Nathan PJ, Newbould RD, Howard J, Miller SR, Bush MA, Hill S, Reiley R, Passchier J, Gunn RN, Matthews PM, Bullmore ET. Pharmacological differentiation of opioid receptor antagonists by molecular and functional imaging of target occupancy and food reward-related brain activation in humans. Mol Psychiatry. 2011 Aug;16(8):826-35, 785. doi: 10.1038/mp.2011.29. Epub 2011 Apr 19. PMID 21502953
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111848 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111848?search=study&search_terms=111848#rs
- Available data/document: Individual Participant Data Set: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register